CLINICAL TRIAL: NCT04062279
Title: Predictors of Parkinson's Disease Progression in Sample of Egyptian Patients; Clinical and Biochemical
Brief Title: Predictors of Parkinson's Disease Progression
Acronym: PDPROG-EGY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ali Shalash, professor, Ain Shams University
Other Study IDs: R58/2018
Record Dates: First submitted 2019-07-02; First posted 2019-08-20 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Cognitive Dysfunction; Biomarkers
Keywords: Parkinson's disease; cognitive dysfunction; alpha synuclein; autoantibodies; progression
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Parkinson Disease 4, Autosomal Dominant Lewy Body; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — blood samples were withdrawn, centrifuged immediately, sera were obtained from collected blood samples, and stored in -20 freezers prior to their collection in Biobank. All collected sera were stored eventually in -80 freezer of the Medical Experimental Research Center (MERC) of Mansoura University
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- case group: patients diagnosed with idiopathic paaarkinson's disease according to the clinical criteria.
  Interventions: Diagnostic Test: serum alpha synuclein autoantibodies, motor and non motor scales

INTERVENTIONS:
Diagnostic Test: serum alpha synuclein autoantibodies, motor and non motor scales — measuring serum alpha synuclein autoantibodies by ELIZA at baseline assessment

SUMMARY:
it is a prospective longitudinal observational study, aiming to to identify clinical, and biochemical baseline predictors of motor and non-motor PD progression in sample of Egyptian patients. it measures the baseline motor, non-motor, biochemical and imaging characteristics at enrollment and its relation to PD progression over 3 years

DETAILED DESCRIPTION:
it is a prospective longitudinal observational study, aiming to to identify clinical, and biochemical baseline predictors of motor and non-motor PD progression in sample of Egyptian patients. it measures the baseline motor, non-motor, biochemical and imaging characteristics at enrollment and its relation to PD progression over 3 years.

The aim of this study is to identify clinical, and biochemical baseline predictors of motor and non-motor PD progression in sample of Egyptian patients.

Methods:

Assessment:-

Time • During the 2 years recruitment of patients from 2019 to 2021, the assessment will be at base line (first clinic visit), after 1yr, and after 2yrs.

Patients will be subjected to:

Clinical assessment:

* At base line, Patients will complete an extensive clinical evaluation, including:

  1. Comprehensive medical history and neurological examination.
  2. Demographic information (sex, age, education level, and occupation), as well as clinical characteristics of them (age at onset, duration of illness, received medications and doses).
  3. Motor assessment; Movement Disorder Society (MDS) -Unified Parkinson's Disease Rating Scale (MDS-UPDRS) he motor portion (Part III) during OFF and ON states, Hoehn & Yahr, and Schwab & England scales.
  4. Gait assessment, Gait will be assessed by:

     Freezing of gait questionnaire Berg balance scale 10 m walk test Timed up and go test

     Physical activity scale for elderly (PASE). Cognitive assessment; MOCA, MMSE. Cognitive assessment : during On state.
* All patients will be evaluated for global cognitive assessment by:
* Mini Mental State Examination (MMSE)Arabic version
* Montreal Cognitive Assessment (MoCA) Arabic version
* The standard battery included cognitive tests in the following domains: visuospatial skills, language, attention, executive functioning, and memory.

  * Visuospatial skills will be assessed by clock drawing test and copy the intersecting pentagons of Addenbrooke's test (Arabic version)
  * Language will be examined by Language similarity & language subset of Addenbrooke's test (Arabic version)
  * Attention will be evaluated by forward &backward digit span tests and by the number of seconds needed to sequence numbers using a pencil (Trail making test A)
  * For the evaluation of memory, participants will complete Wechsler memory subset, and investigators also will use their three-item recall from the MMSE.
  * Executive functions will be measured by Wisconsin card sorting test and also Semantic verbal fluency test .

The non-motor symptoms scales (NMSS). Beck depression inventory (BDI). The Arabic version of The Parkinson's Disease Questionnaire (PDQ-39). Lab investigations MRI brain or CT brain . Serum alpha -Synuclein auto antibodies

All the following will be done at baseline, after 1 year, and after 2 year except, MRI brain and serum alpha-synuclein (only at baseline ).

This study will be approved from the ethical committee of Faculty of Medicine, Ain -Shams University.

ELIGIBILITY:
Inclusion Criteria:

* • All are Arabic-speaking individuals diagnosed with PD by a movement disorder neurologist based on the UK bank criteria for idiopathic Parkinson's disease.

  * An oral informed consent will be taken from the cases before they participate in the study.

Exclusion Criteria:

* Patients with red flag for being diagnosed with IPD and indicating secondary eg: vascular, Neuroleptics or atypical parkinsonism , progressive supranuclear palsy, multiple system atrophy, corticobasal degeneration syndrome, Lewy body dementia

  * Patients with with other comorbid chronic diseases
  * PD patients who refused or could not complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All idiopathic Parkinson patients attending movement disorder clinic meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
predictors of progression of motor features of PD | at 1, 2,3 years follow ups
  change in MDS UPDRS, Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS), from 0 to 260. The MDS-UPDRS has four parts, namely, I: Non-motor Experiences of Daily Living (13 questions) total is from 0 to 52; II: Motor Experiences of Daily Living (13 questions, from 0 to 52) III: Motor Examination (20 questions), total is from 0 to 132; IV: Motor Complications (6 questions, from 0 to 24). In each question: 0=normal; 1=slight; 2= mild; 3=moderate; 4=severe.higher values represent a worse outcome
predictors of progression of non motor features of PD | at 1, 2 ,3 years follow-ups
  changes in Nonmotor, and depression scores.
  Non-Motor Symptom assessment scale for Parkinson's Disease, Symptoms assessed over the last month. Each symptom scored with respect to:
  Severity: from 0 to 3 Frequency: from 1 to 4 Yes/ No answers are not included. score of each question = frequency x severity . There are nine domains: Cardiovascular including falls, Sleep/fatigue, Mood/cognition, Perceptual problems/hallucinations, Attention/memory, Gastrointestinal tract, Urinary, Sexual function, and Miscellaneous. Higher values represent worse outcome.
  Depression assessment scales: Beck depression inventory (BDI) (Higher values represent worse outcome, Arabic version)

SECONDARY OUTCOMES:
development of drug (levodopa) complications | at 1,2, and 3 years
  follow up patients regarding appearance of levodopa related complications using Assessment will be done by Unified Dyskinesia Rating Scale (UDysRS) which is developed to evaluate involuntary movements often associated with treated Parkinson's disease. There are two primary sections: Historical [Part 1 (On-Dyskinesia) and Part 2 (Off-Dystonia)], and Objective [Part 3 (Impairment) and Part 4 (Disability)]
development of gait problems | at1,2, and 3 years
  detecting changes in patients gait. Assessment of gait by Freezing of gait questionnaire (contain 9 questions allocated in 3 parts, score of each question ranges from 0; very mild freezing of gait to 3 or 4 ; with sever freezing of gait), Berg balance scale(to assess the static and dynamic balance by 14 questions with total score =56, each question scored from 0; the sever impairment , to 4 without impairment), 10 meter walk test (individual walks without assistance 10 meters (32.8 feet) and the time is measured, calculate the average of the three trials), and Timed up and go test.
change of quality of life | at 1, 2 ,3 years
  The Arabic version of Parkinson's Disease Questionnaire (PDQ-39), Higher values represent better outcome.

OTHER OUTCOMES:
frequency of dementia and mild cognitive impairment in PD patients | at base line assessment in the first year
  detected by baseline assessment of cognitive functions, using Cognitive scale: Montreal Cognitive Assessment (MoCA) (Arabic version), Visuospatial skills will be assessed by 3-D Wire Cube from Addenbrooke, and Clock Drawing Tests from MoCA test, Language will be examined by semantic fluency Addenbrooke's test (Arabic version), and similarities from IQ Wechsler test, Attention will be evaluated by DIGIT SPAN FROM WECHSLER MEMORY Trail making from MoCA) For the evaluation of memory, participants will complete Wechsler memory subset, and investigators also will use their three-item recall from the Mini-Mental State Examination ( MMSE), Executive functions will be measured by Wisconsin card sorting test and also verbal fluency test from Addenbrooke's test. Higher values represent worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shalash, professor, Principal Investigator — Ain Shams Univeristy
Locations (1):
- Ain Shams Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salama M, Shalash A, Magdy A, Makar M, Roushdy T, Elbalkimy M, Elrassas H, Elkafrawy P, Mohamed W, Abou Donia MB. Tubulin and Tau: Possible targets for diagnosis of Parkinson's and Alzheimer's diseases. PLoS One. 2018 May 9;13(5):e0196436. doi: 10.1371/journal.pone.0196436. eCollection 2018. PMID 29742117
- [Background] Shalash A, Salama M, Makar M, Roushdy T, Elrassas HH, Mohamed W, El-Balkimy M, Abou Donia M. Elevated Serum alpha-Synuclein Autoantibodies in Patients with Parkinson's Disease Relative to Alzheimer's Disease and Controls. Front Neurol. 2017 Dec 22;8:720. doi: 10.3389/fneur.2017.00720. eCollection 2017. PMID 29312137
- [Background] Shalash AS, Hassan DM, Elrassas HH, Salama MM, Mendez-Hernandez E, Salas-Pacheco JM, Arias-Carrion O. Auditory- and Vestibular-Evoked Potentials Correlate with Motor and Non-Motor Features of Parkinson's Disease. Front Neurol. 2017 Feb 27;8:55. doi: 10.3389/fneur.2017.00055. eCollection 2017. PMID 28289399
- [Result] Shalash AS, Hamid E, Elrassas HH, Bedair AS, Abushouk AI, Khamis M, Hashim M, Ahmed NS, Ashour S, Elbalkimy M. Non-Motor Symptoms as Predictors of Quality of Life in Egyptian Patients With Parkinson's Disease: A Cross-Sectional Study Using a Culturally Adapted 39-Item Parkinson's Disease Questionnaire. Front Neurol. 2018 May 24;9:357. doi: 10.3389/fneur.2018.00357. eCollection 2018. PMID 29881368
- [Result] Rosler TW, Salama M, Shalash AS, Khedr EM, El-Tantawy A, Fawi G, El-Motayam A, El-Seidy E, El-Sherif M, El-Gamal M, Moharram M, El-Kattan M, Abdel-Naby M, Ashour S, Muller U, Dempfle A, Kuhlenbaumer G, Hoglinger GU. K-variant BCHE and pesticide exposure: Gene-environment interactions in a case-control study of Parkinson's disease in Egypt. Sci Rep. 2018 Nov 8;8(1):16525. doi: 10.1038/s41598-018-35003-4. PMID 30410011